CLINICAL TRIAL: NCT01622803
Title: Comparison Between Two Methods of Bilateral Stenting for Malignant Hilar Obstruction
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Patients enrollment problem
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kwang Hyuck Lee, Assistant Professor of Medicine, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KH0LEE
Record Dates: First submitted 2012-06-12; First posted 2012-06-19 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Bile Duct Neoplasm; Obstructive Jaundice
MeSH Terms: conditions — Bile Duct Neoplasms; Jaundice, Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- parallel stent (Active Comparator): parallel stent insertion group
  Interventions: Procedure: parallel stent
- Y-stent (Active Comparator): Y-stent insertion group
  Interventions: Device: Y-stent (BONASTENT M-Hilar)

INTERVENTIONS:
Procedure: parallel stent — bilateral parallel stent insertion (right and left side)
  Other Names: bilateral pig tail plastic stent
  Arms: parallel stent
Device: Y-stent (BONASTENT M-Hilar) — Bilateral Y-stent insertion (stent in stent type)
  Other Names: BONASTENT M-Hilar, Standard Sci Tech Inc, Seoul, South Korea
  Arms: Y-stent

SUMMARY:
Internal biliary drainage using stent is used for malignant hilar obstruction such as cholangiocarcinoma, hepatocellular carcinoma and other malignancy including metastasis.

Bilateral drainage is more physiologic and have more long patency than unilateral drainage.

There are two methods of bilateral drainage: Y-stent and side by side.

However there are no clinical data about comparing the effectiveness of these two methods.

Therefore the investigators want to compare the clinical outcomes of two methods:

Y-stent and side by side.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* patient who have obstructive jaundice (bilirubin > 2.0mg/dl) due to hilar malignancy

Exclusion Criteria:

* patients with endoscopic retrograde cholangiogram is not possible
* bleeding tendency (PT INR > 1.5, platelet < 50,000)
* poor general condition (ECOG 3-4) or cardiopulmonary deterioration
* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
The time taken to insert bilateral stent | After the ERCP procedure

CONTACTS AND LOCATIONS:
Overall Officials: Kwang hyuck Lee, MD, phD, Study Director — Division of Gastroenterology, Department of Internal Medicine, Samsung Medical Center, Sungkyunkwan University School of Medicine
Locations (1):
- Samsung Medical Center, Seoul, South Korea